CLINICAL TRIAL: NCT00842712
Title: Open-label, Randomized, Controlled, Multicenter Phase II Trial Investigating 2 Cilengitide Regimens in Combination With Cetuximab and Platinum-based Chemotherapy (Cisplatin/Vinorelbine or Cisplatin/Gemcitabine) Compared to Cetuximab and Platinum-based Chemotherapy Alone as First Line Treatment for Subjects With Advanced NSCLC
Brief Title: Cilengitide and Cetuximab in Combination With Platinum-based Chemotherapy as First-line Treatment for Subjects With Advanced Non Small Cell Lung Cancer (NSCLC)
Acronym: CERTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200037-014; EudraCT Number: 2008-004148-35
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Results first posted 2014-09-30 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: First-line treatment for subjects with advanced NSCLC,; integrin receptor antagonist, EGFR chimerized monoclonal antibody, chemotherapy; safety run-in + randomization part, MTD, PFS, Overall survival time, best overall response
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Metatropic dwarfism | interventions — Cilengitide; Cetuximab; Cisplatin; Gemcitabine; Vinorelbine; Drug Therapy

ARMS (7):
- Safety run-in part: Cil (1000 mg) + Cetuximab + Cis + Gem (Experimental)
  Interventions: Drug: Cilengitide; Drug: Cetuximab; Drug: Cisplatin; Drug: Gemcitabine
- Safety run-in part: Cil (1000 mg) + Cetuximab + Cis + Vin (Experimental)
  Interventions: Drug: Cilengitide; Drug: Cetuximab; Drug: Cisplatin; Drug: Vinorelbine
- Safety run-in part: Cil (2000 mg) + Cetuximab + Cis + Gem (Experimental)
  Interventions: Drug: Cilengitide; Drug: Cetuximab; Drug: Cisplatin; Drug: Gemcitabine
- Safety run-in part: Cil (2000 mg) + Cetuximab + Cis + Vin (Experimental)
  Interventions: Drug: Cilengitide; Drug: Cetuximab; Drug: Cisplatin; Drug: Vinorelbine
- Randomized part: Cil (Once Weekly) + Cetuximab + Chemotherapy (Experimental)
  Interventions: Drug: Cilengitide; Drug: Cetuximab; Drug: Chemotherapy
- Randomized part: Cil (Twice Weekly) + Cetuximab + Chemotherapy (Experimental)
  Interventions: Drug: Cilengitide; Drug: Cetuximab; Drug: Chemotherapy
- Randomized part: Cetuximab + Chemotherapy (Active Comparator)
  Interventions: Drug: Cetuximab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Cilengitide — Cilengitide (Cil) will be administered at a dose of 1000 milligram (mg) as intravenous infusion twice weekly over 1 hour on Days 1 and 4.
  Arms: Safety run-in part: Cil (1000 mg) + Cetuximab + Cis + Gem; Safety run-in part: Cil (1000 mg) + Cetuximab + Cis + Vin
Drug: Cilengitide — Cil will be administered at a dose of 2000 mg as intravenous infusion twice weekly over 1 hour on Days 1 and 4.
  Arms: Safety run-in part: Cil (2000 mg) + Cetuximab + Cis + Gem; Safety run-in part: Cil (2000 mg) + Cetuximab + Cis + Vin
Drug: Cetuximab — Cetuximab will be administered at a dose of 400 milligram per square meter (mg/m^2) as intravenous infusion over 2 hours on Day 1.
  Arms: Safety run-in part: Cil (1000 mg) + Cetuximab + Cis + Gem; Safety run-in part: Cil (1000 mg) + Cetuximab + Cis + Vin; Safety run-in part: Cil (2000 mg) + Cetuximab + Cis + Gem; Safety run-in part: Cil (2000 mg) + Cetuximab + Cis + Vin
Drug: Cisplatin — Cisplatin (Cis) will be administered at a dose of 75 mg/m^2 as intravenous infusion on Day 1.
  Arms: Safety run-in part: Cil (1000 mg) + Cetuximab + Cis + Gem; Safety run-in part: Cil (2000 mg) + Cetuximab + Cis + Gem
Drug: Cisplatin — Cis will be administered at a dose of 80 mg/m^2 as intravenous infusion on Day 1.
  Arms: Safety run-in part: Cil (1000 mg) + Cetuximab + Cis + Vin; Safety run-in part: Cil (2000 mg) + Cetuximab + Cis + Vin
Drug: Gemcitabine — Gemcitabine (Gem) will be administered at a dose of 1250 mg/m^2 as intravenous infusion on Days 1 and 8.
  Arms: Safety run-in part: Cil (1000 mg) + Cetuximab + Cis + Gem; Safety run-in part: Cil (2000 mg) + Cetuximab + Cis + Gem
Drug: Vinorelbine — Vinorelbine (Vin) will be administered at a dose of 25 mg/m^2 as intravenous infusion on Days 1 and 8.
  Arms: Safety run-in part: Cil (1000 mg) + Cetuximab + Cis + Vin; Safety run-in part: Cil (2000 mg) + Cetuximab + Cis + Vin
Drug: Cilengitide — Cil will be administered at a dose of 2000 mg as intravenous infusion once weekly over 1 hour on Days 1, 8 and 15 of each 3-week cycle until progressive disease, death, unacceptable toxicity, or consent withdrawal.
  Arms: Randomized part: Cil (Once Weekly) + Cetuximab + Chemotherapy
Drug: Cilengitide — Cil will be administered at a dose of 2000 mg as intravenous infusion twice weekly over 1 hour on Days 1, 4, 8, 11, 15, and 18 of each 3-week cycle followed by once weekly administration after end of chemotherapy until progressive disease, death, unacceptable toxicity, or consent withdrawal.
  Arms: Randomized part: Cil (Twice Weekly) + Cetuximab + Chemotherapy
Drug: Cetuximab — Cetuximab will be administered at a dose of 400 mg/m^2 as intravenous infusion over 2 hours on Day 1 of Cycle 1 followed by 250 mg/m^2 intravenous infusion over 1 hour once weekly on Days 8 and 15 of Cycle 1 and Days 1, 8, and 15 of all subsequent cycles until progressive disease, death, unacceptable toxicity, or consent withdrawal.
  Arms: Randomized part: Cetuximab + Chemotherapy; Randomized part: Cil (Once Weekly) + Cetuximab + Chemotherapy; Randomized part: Cil (Twice Weekly) + Cetuximab + Chemotherapy
Drug: Chemotherapy — Cis 80 mg/m^2 intravenous infusion on Day 1 + Vin 25 mg/m^2 or Cis 75 mg/m^2 intravenous infusion on Day 1 + Gem 1250 mg/m^2 intravenous infusion on Days 1 and 8 of each 3-week cycle will be administered along with Cil and cetuximab as per Investigator's discretion up to a maximum of 6 cycles.
  Arms: Randomized part: Cetuximab + Chemotherapy; Randomized part: Cil (Once Weekly) + Cetuximab + Chemotherapy; Randomized part: Cil (Twice Weekly) + Cetuximab + Chemotherapy

SUMMARY:
Primary objective of the study's Safety run-in:

- To determine the maximum tolerated dose (MTD) of cilengitide in combination with cetuximab, and platinum-based chemotherapy (cisplatin/vinorelbine or cisplatin/gemcitabine).

Primary objective of the study's Randomization Part:

- To assess the efficacy of cilengitide in combination with cetuximab and platinum-based chemotherapy (cisplatin/vinorelbine or cisplatin/gemcitabine) compared to cetuximab and platinum-based chemotherapy alone in terms of progression-free survival (PFS) time.

Study design and plan:

This is a multicenter, open-label, randomized, controlled Phase II study with a safety run-in part in subjects with advanced non-small cell lung cancer (NSCLC).

During the safety run-in, the regimen was intensified stepwise by cohort (cilengitide intravenous [i.v.] 1000 milligram [mg] to 2000 mg twice a week) in a classical 3+3 subjects (for each platinum-based chemotherapy regimens separately) approach with predefined dose- and schedule reduction rules.

In the safety run-in 12 subjects were included and evaluated for safety and feasibility of different escalating doses of cilengitide administered twice weekly in combination with cetuximab, cisplatin and vinorelbine or gemcitabine.

After completion of the safety run-in, the randomized part will be started, during which all subjects will receive cetuximab and platinum-based chemotherapy (cisplatin/vinorelbine or cisplatin/gemcitabine).

Subjects will be centrally randomized on a 1:1 basis to either Group A or C; Group B will be closed with implementation of Amendment No. 4 (dated 20 December 2010):

• Group A: Cilengitide 2000 mg once weekly (Days 1, 8, and 15 of every 3-week chemotherapy cycle) in combination with cetuximab and platinum-based chemotherapy that will consist of the following:

* Cetuximab once weekly (Days 1, 8, and 15), plus cisplatin on Day 1 and vinorelbine on Days 1 and 8 of every 3-week chemotherapy cycle, or
* Cetuximab once weekly (Days 1, 8, and 15), plus cisplatin on Day 1 and gemcitabine on Days 1 and 8 of every 3-week chemotherapy cycle.

The decision which of the 2 chemotherapy regimens will be applied for a given subject is at the discretion of the treating investigator.

• Group B: Cilengitide 2000 mg twice weekly (Days 1, 4, 8, 11, 15, and 18 of every 3-week chemotherapy cycle) in combination with cetuximab and platinum-based chemotherapy as described for Group A.

Group B will be closed with implementation of Amendment No. 4 (global, dated 20 December 2010). Subjects randomized to Group B before implementation of Amendment No 4 will continue to be treated as planned.

• Group C: Cetuximab and platinum-based chemotherapy as described for Group A

Chemotherapy will be given until radiographically documented progressive disease (PD) or unacceptable toxicity but for no more than 6 cycles.

Cilengitide and cetuximab will be given until radiographically documented PD or unacceptable toxicity.

Randomization will be performed centrally using an interactive voice/web response system (IXRS). A stratified block randomization procedure will be employed using chosen first-line chemotherapy (cisplatin/vinorelbine versus cisplatin/gemcitabine) as stratification criterion.

DETAILED DESCRIPTION:
Schedule of visits and assessments:

Pre-screening Visit (Within 2 weeks prior to screening):

In an initial step subjects with newly diagnosed NSCLC (suspected or already established diagnosis) will be offered to have their tumor assessed locally for Epidermal Growth Factor Receptor (EGFR) expression. After giving specific written informed consent to this analysis, they will be formally registered and the tissue will be analyzed.

Signing of informed consent for local immunohistochemistry (IHC) based EGFR expression determination; EGFR expression testing in local pathology laboratory using archived tumor material; Demographics, that is, subject initial, date of birth, gender, ethnicity/race, height; Allocation of subject number; Date of initial diagnosis; Tumor characteristics (histology, localization, metastasis, Tumor-Nodes-Metastases (TNM) classification).

Screening Visit (Within 3 weeks prior to randomization):

Signing of informed consent for study participation (only if pre-screening positive and with an EGFR expression >=200); Archived tumor material for biomarker analysis including EGFR, k-ras, b-raf, pathology and possible additional biomarker research including mutation testing; Relevant medical history; Prior treatment of underlying tumor; Physical examination including vital signs (including body weight, without body surface area [BSA]); ECOG-performance status; Central 12-lead electrocardiogram (ECG); Pulmonary function test; Baseline imaging within 4 weeks prior to randomization (RECIST): At least chest + abdomen computed tomography (CT) (or magnetic resonance imaging [MRI] if there are contraindications to CT); Documentation of concomitant medications and adverse events (AEs); Safety laboratory assessments (hematology including coagulation parameters and biochemistry); Blood sampling for Human anti-chimeric antibody (HACA) assessment; Serum pregnancy test for women of childbearing potential within 7 days to the start of study medication; In-/exclusion criteria review; Randomization, (to be performed <=7 days before start of therapy); Optional: additional written informed consent for pharmacogenetics testing and optional: blood sampling for pharmacogenetics testing (only applicable for randomized study part).

Day 1 of Each Cycle (Start of Cycle Visit) (At start of each chemotherapy cycle) Before start of first cycle: randomization should be performed <=7 days before start of therapy; Physical examination including vital signs (including body weight and BSA); Assessment of cardiovascular specific symptoms; Documentation of AEs; Concomitant medication; Safety laboratory assessments (hematology including coagulation parameters and biochemistry) must be available before start of chemotherapy; Central Holter ECG before start of treatment until the end of infusion of cilengitide (for Group C subjects until the 1 hour after the end of infusion of cetuximab) on Day 1 of the first cycle only; Central standard ECG Cycles 2-6; ECOG-performance status; Administration of cilengitide (Groups A and B); Administration of cetuximab (all subjects); Administration of cisplatin/vinorelbine or cisplatin/gemcitabine (all subjects; first 6 cycles only); Blood sampling for plasma circulating markers (only on Day 1 of Cycle 1 at pre-dose and at the end of the cisplatin infusion); Additional blood sampling for Common Toxicity Criteria (CTC)/circulating endothelial cell (CEC) assessment (only pre-dose on Day 1 of Cycle 1 and Cycle 2); Blood sampling for cilengitide pharmacokinetic (PK) (6-10 subjects of Group B only; Cycle 1 only; see Section 7.4.1 for details) (at dedicated sites only); Blood sampling for cetuximab PK (all subjects of Group A only; Cycles 1 and 2 only); Blood sampling for vinorelbine PK (6-10 subjects of Groups B and C; Cycle 1 only) (at dedicated sites only).

Days 4, 11 and 18

Days 4, 11, and 18 of Each Cycle (Group B only) Vital signs (without BSA/body weight); Administration of cilengitide.

Days 4 and 11 (additional examinations during the first 2 weeks of first cycle of safety run-in): safety laboratory assessments (hematology including coagulation parameters and biochemistry).

Days 8 and 15

Days 8 and 15 of Each Cycle: Vital signs (without BSA/weight); assessment of cardiovascular specific symptoms; documentation of AEs; concomitant medication; administration of cilengitide (Groups A and B); administration of cetuximab; administration of vinorelbine or gemcitabine (all subjects; Day 8 of the first 6 cycles only); blood sampling for pro-brain natriuretic peptide (proBNP) (Cycle 1 Day 8 only); blood sampling for cetuximab PK (all subjects of Group A only; Days 8 and 15 of Cycle 1 and Day 8 of Cycle 2 only); blood sampling for plasma circulating markers (all subjects; Days 8 and 15 of first cycle only at pre dose, for each subsequent cycle on Day 8 only).

Days 8 and 15 (additional examinations during safety run-in): safety laboratory assessments (hematology including coagulation parameters and biochemistry) must be available before start of chemotherapy.

Once weekly safety lab evaluation during safety run-in (after end of chemotherapy): safety laboratory assessments (hematology including coagulation parameters and biochemistry).

6-weekly Evaluation Visit (Every 6 weeks +/- 2 days after randomization until final tumor assessment (FTA) visit): Physical examination including vital signs (without BSA/weight); assessment of cardiovascular specific symptoms; documentation of AEs; concomitant medication; ECOG-performance status; central standard ECG after cycle 6 only; CT scan or MRI; safety laboratory assessments (hematology including coagulation parameters and biochemistry); serum pregnancy test for women of childbearing potential. Blood sampling for plasma circulating markers during maintenance treatment only, and for CTC/CEC (only once after 6 cycles of chemotherapy).

Final Tumor Assessment Visit (At occurrence of PD and/or before start of any other systemic anti-tumor therapy): Physical examination including vital signs (without BSA); documentation of AEs; concomitant medication; ECOG-performance status; CT scan or MRI; safety laboratory assessments (hematology including coagulation parameters and biochemistry); blood sampling for plasma circulating markers and CTC/CEC; serum pregnancy test.

End-of-Study (EoS) Visit (Around 28 days after the last investigational medicinal product [cilengitide or cetuximab] administration, or before other anticancer treatment starts, but not before the FTA visit): Physical examination including vital signs (without BSA); documentation of AEs. If a subject begins a subsequent anticancer therapy, the AE reporting period for non-serious AEs will end at the time the new treatment starts; ECOG-performance status; concomitant medication; safety laboratory assessments (hematology including coagulation parameters and biochemistry); blood sampling for HACA assessment; central 12-lead ECG; reason for discontinuation.

Survival Follow-up (Every 2 months after EoS visit): Each subject's survival status and any further anti-cancer treatments will be documented every 2 months after the end of study visit until death, loss to follow-up, or consent withdrawal.

All subjects will be treated with platinum-based chemotherapy for a maximum of 6 cycles (that is, 18 weeks), until PD or death, unacceptable toxicity, or until the subject withdraws consent. Subjects who do not experience PD after 6 cycles of platinum-based treatment will continue treatment with cilengitide (Groups A and B) and cetuximab (Group A, B and C). Subjects who discontinue treatment without PD will remain on study. Response assessment will continue every 6 weeks until PD or until other anti-tumor treatment is started. Upon this occurrence, all study medication should be discontinued and a final tumor assessment (FTA) visit will be carried out. The end-of-study visit should be performed around 4 weeks after the last investigational medicinal product administration but not before the FTA visit.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent obtained before undergoing any study-related activities.
2. Male or female, at least 18 years of age
3. Histologically confirmed NSCLC, Stage IIIb with documented malignant pleural effusion or Stage IV (according to staging system 6th edition)
4. EGFR expression greater than or equal to (>=) 200 on tumor tissue determined by local testing using the kit and testing procedures described in the study Manual of Operations (MOP)
5. Archived tumor material sample for central histology and further biomarker research including mutational analysis of genes such as EGFR, k-ras, b-raf (material details described in the study MOP)
6. At least 1 radiographically documented measurable lesion in a previously non-irradiated area according to evaluation criteria in solid tumors (RECIST), i.e. this lesion must be adequately measurable in at least 1 dimension (longest diameter [LD] to be recorded) as >=2 centimeter (cm) by conventional techniques or ≥1 cm by spiral CT scan
7. Eastern Cooperative Oncology Group (ECOG)-performance status 0-1
8. Leukocyte count >=3.0 x 10^9 per liter (/L)
9. Absolute neutrophil count (ANC) >=1.5 x 10^9/L
10. Platelets >=100 x 10^9/L
11. Hemoglobin >=9 gram per deciliter (g/dL) (without transfusions)
12. Bilirubin less than or equal to (<=) 1.5 x upper limit of normality (ULN)
13. Aspartate Aminotransferase (AST) <=5 x ULN and Alanine Aminotransferase (ALT) <=5 x ULN
14. Serum creatinine <=1.25 x ULN and/or creatinine clearance >=60 milliliter per minute (mL/min)
15. Prothrombin time (PT), international normalized ratio (INR) within normal limits and partial thromboplastin time (PTT) below upper limit of normal.
16. Sodium and potassium within normal limits or <=10% above or below (supplementation permitted).
17. Effective contraception for both male and female subjects (if the risk of conception exists). If female, she must: be neither pregnant nor breast-feeding, nor attempting to conceive, use a highly effective method of contraception for at least 7 days before entry into the trial, throughout the entire duration of the trial and for 6 months following completion of the last dose of trial medication. A highly effective method of contraception is defined as those which result in a low failure rate (that is, <1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, intrauterine devices (IUDs) (hormonal or copper-based), sexual abstinence or vasectomized partner, or be post-menopausal or surgically sterilized. If male, he must be willing to use contraception to avoid pregnancies for at least 7 days before entry into the trial, throughout the entire duration of the trial and for 6 months following the last dose of trial medication. Two negative semen analyses post-vasectomy have to be available in order to be considered infertile

Exclusion criteria:

1. Prior treatment with an antibody or molecule targeting EGFR- and/or vascular endothelial growth factor receptor (VEGFR)-related signaling pathways
2. Previous chemotherapy for NSCLC including prior adjuvant therapy
3. History of or current brain metastasis and/or leptomeningeal disease (known or suspected)
4. Radiotherapy (except localized radiotherapy for pain relief), major surgery or any intake of investigational drug in the 30 days before the start of study treatment entry
5. Concurrent chronic immunosuppressive or hormone anti-cancer therapy (physiologic hormone replacement or corticosteroid treatment for chronic obstructive pulmonary disease [COPD] is allowed)
6. Clinically relevant coronary artery disease (New York Heart Association [NYHA] functional angina classification III/IV), congestive heart failure (NYHA III/IV), clinically relevant cardiomyopathy, history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia
7. History of coagulation disorder associated with bleeding, recurrent or recent thrombotic events or history of hemoptysis related to bronchopulmonary cancer. Hemoptysis is defined as coughing more than a teaspoon of red blood per day
8. Recent peptic ulcer disease (endoscopically proven gastric, duodenal or esophageal ulcer) within 6 months of study treatment start
9. Presence of any contra-indication to treatment with cilengitide, cetuximab, cisplatin and vinorelbine or gemcitabine including:

   * Known hypersensitivity to cilengitide, cetuximab, cisplatin, vinorelbine, or gemcitabine or to any of the excipients of these drugs
   * Superior vena cava syndrome contra-indicating hydration
   * Symptomatic peripheral neuropathy National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grade >=2 and/or ototoxicity NCI CTC AE Grade >=2, except if due to trauma or mechanical impairment due to tumor mass
   * Phenytoin (introduced to prevent the anticonvulsant effect of certain anticancer drugs) (contra-indication for cisplatin)
   * Yellow Fever Vaccine, Live Attenuated Vaccines (contra-indications for cisplatin)
10. Pregnancy or lactation period
11. Concurrent treatment with a non-permitted drug
12. Treatment with any other investigational product within the past 30 days
13. Previous malignancy other than NSCLC in the last 5 years except for basal cell cancer of the skin or pre-invasive cancer of the cervix
14. Medical or psychological conditions that would not permit the subject to complete the study or sign informed consent
15. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such
16. Patients with hepatitis, massive liver metastases (>75%), current alcoholism or liver cirrhosis (because of vinorelbine and gemcitabine)
17. Patients who have been therapeutically anticoagulated
18. Legal incapacity or limited legal capacity
19. Significant disease (for example, interstitial lung disease) which, in the investigator's opinion, would exclude the subject from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2009-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (44):
- Belgium (6):
  - Research Site, Antwerpen (Edegem)
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Gosselies
  - Research Site, Leuven
  - Research Site, Mons
- Czechia (2):
  - Research Site, Liberec
  - Research Site, Usti Nach Labem
- France (10):
  - Research Site, Bobigny
  - Research Site, Bordeaux
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nantes - Saint Herblain
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Vandœuvre-lès-Nancy
- Germany (14):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Darmstadt
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Goch
  - Research Site, Halle-Dölau
  - Research Site, Hamburg
  - Research Site, Lübeck
  - Research Site, Mannheim
  - Research Site, Munich
  - Research Site, Offenbach
  - Research Site, Oldenburg
  - Research Site, Wiesbaden
- Research Site, Dublin, Ireland
- Italy (4):
  - Research Site, Avellino
  - Research Site, Bologna
  - Research Site, Meldola
  - Research Site, Rome
- Poland (5):
  - Research Site, Lublin
  - Research Site, Otwock
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wodzisław Śląski
- Spain (2):
  - Research Site, Baracaldo Vizcaya
  - Research Site, Barcelona

REFERENCES:
- [Derived] Vansteenkiste J, Barlesi F, Waller CF, Bennouna J, Gridelli C, Goekkurt E, Verhoeven D, Szczesna A, Feurer M, Milanowski J, Germonpre P, Lena H, Atanackovic D, Krzakowski M, Hicking C, Straub J, Picard M, Schuette W, O'Byrne K. Cilengitide combined with cetuximab and platinum-based chemotherapy as first-line treatment in advanced non-small-cell lung cancer (NSCLC) patients: results of an open-label, randomized, controlled phase II study (CERTO). Ann Oncol. 2015 Aug;26(8):1734-40. doi: 10.1093/annonc/mdv219. Epub 2015 May 4. PMID 25939894

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): Feb 2009/Jun 2012. Clinical data cut-off: 26 Jun 2013, Study completion date: July 2013.
Pre-assignment Details: In safety run-in part of study, a total of 12 participants were enrolled and treated. In randomized part of study, 220 participants were enrolled and out of these 220 participants, 215 were treated.
Groups:
- Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Gem: Cilengitide (Cil) 1000 milligram (mg) intravenous infusion twice weekly over 1 hour on Days 1 and 4 + Cetuximab 400 milligram per square meter (mg/m^2) intravenous infusion over 2 hours on Day 1 + Cisplatin (Cis) 75 mg/m^2 intravenous infusion on Day 1 + Gemcitabine (Gem) 1250 mg/m^2 intravenous infusion on Days 1 and 8 for 3 weeks.
- Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Vin: Cil 1000 mg intravenous infusion twice weekly over 1 hour on Days 1 and 4 + Cetuximab 400 mg/m^2 intravenous infusion over 2 hours on Day 1 + Cis 80 mg/m^2 intravenous infusion on Day 1 + Vinorelbine (Vin) 25 mg/m^2 intravenous infusion on Days 1 and 8 for 3 weeks.
- Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Gem: Cil 2000 mg intravenous infusion twice weekly over 1 hour on Days 1 and 4 + Cetuximab 400 mg/m^2 intravenous infusion over 2 hours on Day 1 + Cis 75 mg/m^2 intravenous infusion on Day 1 + Gem 1250 mg/m^2 intravenous infusion on Days 1 and 8 for 3 weeks.
- Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Vin: Cil 2000 mg intravenous infusion twice weekly over 1 hour on Days 1 and 4 + Cetuximab 400 mg/m^2 intravenous infusion over 2 hours on Day 1 + Cis 80 mg/m^2 intravenous infusion on Day 1 + Vin 25 mg/m^2 intravenous infusion on Days 1 and 8 for 3 weeks.
- Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy: Cil 2000 mg intravenous infusion once weekly over 1 hour on Days 1, 8 and 15 of each 3-week cycle + Cetuximab 400 mg/m^2 intravenous infusion over 2 hours on Day 1 of Cycle 1 followed by cetuximab 250 mg/m^2 intravenous infusion over 1 hour once weekly on Days 8 and 15 of Cycle 1 and Days 1, 8, and 15 of all subsequent cycles until progressive disease, death, unacceptable toxicity, or consent withdrawal. Chemotherapy (Cis 80 mg/m^2 intravenous infusion on Day 1 + Vin 25 mg/m^2 or Cis 75 mg/m^2 intravenous infusion on Day 1 + Gem 1250 mg/m^2 intravenous infusion on Days 1 and 8 of each 3-week cycle) was administered along with Cil and cetuximab as per Investigator's discretion up to a maximum of 6 cycles.
- Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy: Cil 2000 mg intravenous infusion twice weekly over 1 hour on Days 1, 4, 8, 11, 15, and 18 of each 3-week cycle followed by once weekly administration after end of chemotherapy + Cetuximab 400 mg/m^2 intravenous infusion over 2 hours on Day 1 of Cycle 1 followed by cetuximab 250 mg/m^2 intravenous infusion over 1 hour once weekly on Days 8 and 15 of Cycle 1 and Days 1, 8, and 15 of all subsequent cycles until progressive disease, death, unacceptable toxicity, or consent withdrawal. Chemotherapy (Cis 80 mg/m^2 intravenous infusion on Day 1 + Vin 25 mg/m^2 or Cis 75 mg/m^2 intravenous infusion on Day 1 + Gem 1250 mg/m^2 intravenous infusion on Days 1 and 8 of each 3-week cycle) was administered along with Cil and cetuximab as per Investigator's discretion up to a maximum of 6 cycles.
- Randomized Part: Cetuximab + Chemotherapy: Cetuximab 400 mg/m^2 intravenous infusion over 2 hours on Day 1 of Cycle 1 followed by cetuximab 250 mg/m^2 intravenous infusion over 1 hour once weekly on Days 8 and 15 of Cycle 1 and Days 1, 8, and 15 of all subsequent cycles until progressive disease, death, unacceptable toxicity, or consent withdrawal. Chemotherapy (Cis 80 mg/m^2 intravenous infusion on Day 1 + Vin 25 mg/m^2 or Cis 75 mg/m^2 intravenous infusion on Day 1 + Gem 1250 mg/m^2 intravenous infusion on Days 1 and 8 of each 3-week cycle) was administered along with Cil and cetuximab as per Investigator's discretion up to a maximum of 6 cycles.
Period: Safety Run-in Part
Arm/Group | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Gem | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Vin | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Gem | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Vin | Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cetuximab + Chemotherapy
Started | 3 | 3 | 3 | 3 | 0 | 0 | 0
Completed | 0 | 1 | 3 | 2 | 0 | 0 | 0
Not Completed | 3 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 3 | 1 | 0 | 1 | 0 | 0 | 0
Period: Randomized Part
Arm/Group | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Gem | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Vin | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Gem | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Vin | Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cetuximab + Chemotherapy
Started | 0 | 0 | 0 | 0 | 85 | 51 | 84
Treated | 0 | 0 | 0 | 0 | 85 | 50 | 80
Completed | 0 | 0 | 0 | 0 | 85 | 50 | 78
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 6
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 0 | 1 | 4
Not completed — Ongoing at cut-off date | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized to trial treatment.
Groups:
- Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Gem: Cil 1000 mg intravenous infusion twice weekly over 1 hour on Days 1 and 4 + Cetuximab 400 mg/m^2 intravenous infusion over 2 hours on Day 1 + Cis 75 mg/m^2 intravenous infusion on Day 1 + Gem 1250 mg/m^2 intravenous infusion on Days 1 and 8 for 3 weeks.
- Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Vin: Cil 1000 mg intravenous infusion twice weekly over 1 hour on Days 1 and 4 + Cetuximab 400 mg/m^2 intravenous infusion over 2 hours on Day 1 + Cis 80 mg/m^2 intravenous infusion on Day 1 + Vin 25 mg/m^2 intravenous infusion on Days 1 and 8 for 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Gem | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Vin | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Gem | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Vin | Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cetuximab + Chemotherapy | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 85 | 51 | 84 | 232
Age, Customized [Number; unit: participants]
  Less than 65 years | 3 | 2 | 3 | 3 | 68 | 37 | 66 | 182
  Greater than or equal to 65 years | 0 | 1 | 0 | 0 | 17 | 14 | 18 | 50
Gender [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 2 | 34 | 19 | 27 | 85
  Male | 2 | 3 | 1 | 1 | 51 | 32 | 57 | 147

OUTCOME MEASURES:

1. Primary Outcome: Safety run-in Part: Number of Participants With Dose Limiting Toxicities (DLTs)
Time Frame: Up to Week 3
Population: DLT population included all participants who completed first 3 weeks of treatment (first chemotherapy cycle) or who discontinued treatment due to any DLT during the first 3 weeks of treatment in the safety-run-in part.
Measure: Number; unit: participants
Groups:
- Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Gem: Cil 1000 mg intravenous infusion twice weekly over 1 hour on Days 1 and 4 + Cetuximab 400 milligram per square meter (mg/m^2) intravenous infusion over 2 hours on Day 1 + Cis 75 mg/m^2 intravenous infusion on Day 1 + Gem 1250 mg/m^2 intravenous infusion on Days 1 and 8 for 3 weeks.
Arm/Group | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Gem | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Vin | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Gem | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Vin
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 0 | 0 | 0 | 0

2. Primary Outcome: Randomized Part: Progression Free Survival (PFS) Time - Independent Read
Description: The PFS time is defined as the duration from randomization to either first observation of progressive disease (PD) or occurrence of death due to any cause. Independent Read is the assessment of all imaging centrally by an Independent Review Committee (IRC).
Time Frame: Time from randomization until disease progression, death or last tumor assessment, reported between day of first participant randomized, that is, Feb 2009 until cut-off date, (26 Jun 2013)
Population: Intent-to-treat (ITT) population included all participants who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cetuximab + Chemotherapy
Number analyzed (Participants) | 85 | 51 | 84
months | 6.2 [5.6 to 7.4] | 5.6 [4.0 to 7.5] | 5.0 [4.2 to 5.6]
Statistical Analysis 1: Comparison: Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy vs Randomized Part: Cetuximab + Chemotherapy; PFS Time: Independent read; Test type: Superiority or Other; p = 0.0845, Log Rank; Hazard Ratio (HR) = 0.718, 95% CI 2-sided [0.492 to 1.048]

3. Secondary Outcome: Randomized Part: Progression Free Survival (PFS) Time - Investigator Read
Description: The PFS time is defined as the duration from randomization to either first observation of progressive disease (PD) or occurrence of death due to any cause. Investigator read is the assessment of all imaging by the treating physician at the local trial site.
Time Frame: as for outcome 2
Population: ITT population included all participants who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cetuximab + Chemotherapy
Number analyzed (Participants) | 85 | 51 | 84
months | 5.6 [5.4 to 6.7] | 5.6 [4.2 to 7.0] | 5.3 [4.2 to 5.7]
Statistical Analysis 1: Comparison: Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy vs Randomized Part: Cetuximab + Chemotherapy; Test type: Superiority or Other; p = 0.5912, Log Rank; Hazard Ratio (HR) = 0.909, 95% CI 2-sided [0.642 to 1.286]

4. Secondary Outcome: Randomized Part: Overall Survival (OS) Time
Description: The OS time is defined as the time (in months) from randomization to death or last day known to be alive. Participants without event are censored at the last date known to be alive or at the clinical cut-off date, whatever is earlier.
Time Frame: Time from randomization until death or last day known to be alive, reported between day of first participant randomized, that is, Feb 2009 until cut-off date,(26 Jun 2013)
Population: ITT population included all participants who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cetuximab + Chemotherapy
Number analyzed (Participants) | 85 | 51 | 84
months | 13.6 [9.5 to 18.6] | 13.6 [8.7 to 16.7] | 9.7 [7.9 to 13.4]
Statistical Analysis 1: Comparison: Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy vs Randomized Part: Cetuximab + Chemotherapy; Test type: Superiority or Other; p = 0.2648, Log Rank; Hazard Ratio (HR) = 0.813, 95% CI 2-sided [0.564 to 1.171]

5. Secondary Outcome: Randomized Part: Best Overall Response (BOR) Rate
Description: The BOR rate is defined as the percentage of participants having achieved confirmed complete response (CR) or partial response (PR) as the best overall response, based on radiological assessments (based on response evaluation criteria in solid tumors [RECIST]) as assessed by Independent Review Committee (IRC): CR = disappearance of all target lesions; PR = at least 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Time from randomization until disease progression, death or last tumor assessment, reported between day of first participant randomized, that is, Feb 2009 until cut-off date,(26 Jun 2013)
Population: ITT population included all participants who were randomized to trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cetuximab + Chemotherapy
Number analyzed (Participants) | 85 | 51 | 84
percentage of participants | 37.6 [27.4 to 48.8] | 27.5 [15.9 to 41.7] | 29.8 [20.3 to 40.7]

6. Secondary Outcome: Randomized Part: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from first administration of trial treatment until the date of the first occurrence of one of the events defining treatment failure: Progressive Disease (PD) assessed by the investigator, discontinuation of treatment due to PD, discontinuation of treatment due to an adverse event (AE), start of any new anticancer therapy, or withdrawal of consent or death within 60 days of the last tumor assessment or first administration of trial treatment. Time to treatment failure was assessed according to modified World Health Organization (WHO) criteria by Independent Review Committee (IRC).
Time Frame: Time from randomization until treatment failure or last tumor assessment, reported between day of first participant randomized, that is, Feb 2009 until cut-off date,(26 Jun 2013)
Population: ITT population included all participants who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cetuximab + Chemotherapy
Number analyzed (Participants) | 85 | 51 | 84
months | 4.4 [3.5 to 5.6] | 2.8 [1.4 to 4.2] | 4.2 [2.8 to 5.3]

ADVERSE EVENTS:
Time Frame: Time from first dose up to 28 days after last dose of study treatment, reported between day of first participant randomized, that is, Feb 2009 until cut-off date (26 Jun 2013)
Description: The analysis was performed on safety population, defined as all participants who received any dose of the trial treatment (cilengitide, cetuximab, or chemotherapy), whereby participants were analyzed according to the actual treatment they received.
Arm/Group | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Gem | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Vin | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Gem | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Vin | Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy | Randomized Part: Cetuximab + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 1/3 | 0/3 | 42/85 | 29/50 | 45/80
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 84/85 | 48/50 | 78/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Gem (N=3) | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Vin (N=3) | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Gem (N=3) | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Vin (N=3) | Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy (N=85) | Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy (N=50) | Randomized Part: Cetuximab + Chemotherapy (N=80)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 5 | 8
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 3
PYREXIA (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1
ASTHENIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
DISEASE PROGRESSION (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
MALAISE (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
IMPAIRED HEALING (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MEDICAL DEVICE COMPLICATION (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 4
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CYSTITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
LUNG INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
NAIL BED INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
PROTEUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 4
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
PROCTITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
AORTIC THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
ARTERIAL DISORDER (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
AXILLARY VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
PERIPHERAL EMBOLISM (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SHOCK (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
VENA CAVA THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
CONVULSION (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
COMA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
STATUS EPILEPTICUS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
FAILURE TO ANASTOMOSE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
STRESS CARDIOMYOPATHY (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
TUMOUR EMBOLISM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOACUSIS (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PERIORBITAL OEDEMA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Gem (N=3) | Safety run-in Part: Cil (1000 mg) + Cetuximab + Cis + Vin (N=3) | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Gem (N=3) | Safety run-in Part: Cil (2000 mg) + Cetuximab + Cis + Vin (N=3) | Randomized Part: Cil (Once Weekly) + Cetuximab + Chemotherapy (N=85) | Randomized Part: Cil (Twice Weekly) + Cetuximab + Chemotherapy (N=50) | Randomized Part: Cetuximab + Chemotherapy (N=80)
RASH (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 3 | 35 | 17 | 29
ACNE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 19 | 11 | 17
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 17 | 7 | 16
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 13 | 7 | 9
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 13 | 5 | 9
SKIN TOXICITY (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 10 | 8 | 7
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 7 | 6 | 3
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 6 | 2 | 6
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 4
NAIL TOXICITY (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 3 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 49 | 26 | 42
DIARRHOEA (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 21 | 13 | 22
VOMITING (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 17 | 13 | 22
CONSTIPATION (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 17 | 14 | 19
STOMATITIS (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 15 | 10 | 11
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 7 | 5 | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 7 | 1 | 6
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 4 | 5 | 2
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
FATIGUE (General disorders) | 3 | 3 | 1 | 1 | 29 | 13 | 19
ASTHENIA (General disorders) | 0 | 0 | 0 | 0 | 20 | 14 | 22
PYREXIA (General disorders) | 1 | 0 | 0 | 0 | 7 | 13 | 14
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0 | 0 | 5 | 5 | 5
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 5 | 5 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 0 | 0 | 5 | 2 | 2
CHILLS (General disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 2
XEROSIS (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 42 | 21 | 34
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 33 | 21 | 22
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 28 | 16 | 21
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 20 | 7 | 9
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 4 | 3 | 4
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 4 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 30 | 13 | 21
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 18 | 9 | 7
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 10 | 5 | 7
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 6 | 3 | 6
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 6 | 1 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 13 | 11 | 12
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 0 | 10 | 9 | 13
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 9 | 10 | 7
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 11 | 6 | 5
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 7
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 5
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 5
WEIGHT DECREASED (Investigations) | 0 | 0 | 1 | 0 | 9 | 3 | 15
HAEMOGLOBIN DECREASED (Investigations) | 0 | 3 | 0 | 1 | 8 | 7 | 7
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 3 | 5 | 5
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 3 | 0 | 0 | 6 | 1 | 3
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 5 | 0 | 4
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 6 | 1 | 1
HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0 | 9 | 6 | 6
DYSGEUSIA (Nervous system disorders) | 1 | 0 | 1 | 0 | 7 | 4 | 5
DIZZINESS (Nervous system disorders) | 2 | 0 | 1 | 1 | 8 | 4 | 2
PARAESTHESIA (Nervous system disorders) | 0 | 3 | 0 | 0 | 3 | 1 | 8
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 3 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 13 | 8 | 7
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 10 | 3 | 6
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 3 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 5
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 4
PARONYCHIA (Infections and infestations) | 1 | 0 | 1 | 0 | 14 | 1 | 8
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 2 | 0 | 5 | 5 | 7
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 5 | 5
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 2 | 5
ANXIETY (Psychiatric disorders) | 0 | 0 | 0 | 0 | 4 | 4 | 8
INSOMNIA (Psychiatric disorders) | 1 | 0 | 0 | 1 | 4 | 3 | 9
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 4
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 9 | 6 | 5
HYPOTENSION (Vascular disorders) | 0 | 1 | 0 | 1 | 1 | 4 | 4
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 0 | 10 | 7 | 5
DYSURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 4 | 4 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
TINNITUS (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 6
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1
HIRSUTISM (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 1
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0
INTERTRIGO (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4 | 1 | 0
ERUCTATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ORAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
OROPHARYNGEALPAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 3 | 1 | 1
MIGRAINE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ANOREXIA (Metabolism and nutrition disorders) | 2 | 3 | 1 | 1 | 0 | 0 | 0
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
IRON OVERLOAD (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 0 | 4 | 1 | 0
PERIPHERAL COLDNESS (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
THROMBOPHLEBITIS (Vascular disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 1
CATHETER SITE INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
NAIL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 4 | 0 | 0
RHINITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 2
TRACHEOBRONCHITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
VAGINAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 2 | 0 | 0 | 2 | 0 | 2
PLATELET COUNT DECREASED (Investigations) | 0 | 2 | 0 | 0 | 5 | 1 | 3
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 3
BLOOD CREATINE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
BLOOD SODIUM DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 2
VISION BLURRED (Eye disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1
BLEPHARITIS (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
EYE IRRITATION (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
EYE PAIN (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 3 | 0 | 3
LEUKOCYTURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
POLYURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
BRADYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 1 | 3 | 2 | 1
DYSPAREUNIA (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days